CLINICAL TRIAL: NCT03501394
Title: What Are the Factors Affecting Neoadjuvant Chemotherapy Efficacy in Breast Cancer? A Non-invasive in Vivo Study Using Specialist Magnetic Resonance (MR) Methods
Brief Title: What Factors Affect Breast Cancer Neoadjuvant Chemotherapy Efficacy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2/108/7; 234794 (Other: Integrated Research Approval System project ID); 17/LO/1777 (Other: Research Ethics Committee Reference)
Record Dates: First submitted 2018-03-28; First posted 2018-04-18 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Breast Neoplasm Malignant Breast Tissue
Keywords: Magnetic Resonance Imaging; Neoadjuvant Chemotherapy
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Patient Health Questionnaire

STUDY DESIGN:
Intervention Model Description: Single group longitudinal study.
Masking Description: Single group with one arm and no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): 25 patients with pathologically confirmed invasive breast cancer who will undergo neoadjuvant chemotherapy treatment (NACT) and surgery will be recruited. During the study, patients will receive the standard care and the current study will not alter the care plan offered to them. All patients in the single arm will undergo 4 magnetic resonance imaging scan sessions. Histopathological analysis will be performed on the core biopsy and tumour tissue removed in surgery. Health questionnaire will be completed by each patient.
  Interventions: Other: Magnetic Resonance Imaging; Other: Histopathological Analysis; Other: Health Questionnaire

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Patients will undergo 4 MRI sessions during NACT treatment. The first scan will take place at treatment baseline before their first cycle of NACT treatment. The second scan will take place following the first treatment cycle prior to the second treatment cycle. Likewise, the third and last scan will take place after the third treatment cycle and sixth (final) treatment cycle prior to surgery. MRI scan sessions will be composed of research scans including diffusion and lipid profiling MR imaging methods and MR spectroscopy (MRS) methods.
Other: Histopathological Analysis — Study specific analysis will be performed on the core biopsy and tissue removed in surgery following the completion of NACT treatment. Standard routine histological analysis will be performed, as well as study specific analysis for immunostaining, grading and slide scan imaging for measurement of cellularity markers.
Other: Health Questionnaire — Health and demographic information will be collected.

SUMMARY:
Breast cancer is the most prevalent cancer affecting women. To treat locally advanced breast cancers, neoadjuvant chemotherapy (NACT) is often carried out before surgery to reduce the tumour size to allow breast conservation surgery. However, treatment response for individual patients varies, where the tumour may not respond to treatment and the quality of patient care is compromised if the NACT treatment plan is not optimised. Therefore, the assessment of NACT efficacy is beneficial for the early identification of these patients and appropriate management of treatment.

Breast tumours have unique features compared to healthy tissue, including abnormal tissue structure and biochemical composition. With NACT there are specific changes to such tumour features indicating tumour treatment response.

The purpose of this study is to establish how the changes to breast tumour features following NACT treatment are seen in non-invasive imaging. This study will look at scans of breast tumours using magnetic resonance imaging (MRI). Changes to tissue structure will be measured by advanced diffusion MRI techniques and changes to tumour related biochemical substances will be measured by advanced magnetic resonance spectroscopy techniques. The investigators aim to assess if these techniques can provide information on the tumour treatment response following subsequent rounds of NACT treatment.

In this longitudinal study, 25 patients undergoing NACT will be recruited for four repeated MRI investigations over the course of NACT treatment. Magnetic resonance (MR) measurements of tissue microstructure and biochemical composition will be compared against histological measurements and radiological assessments of treatment response.

The study will recruit patients undergoing treatment at the NHS Grampian. This research is funded by Friends of ANCHOR, Tenovus Scotland Grampian and the NHS Grampian Endowment Research Fund.

DETAILED DESCRIPTION:
In this single group longitudinal study, the investigators propose that functional images from magnetic resonance (MR) methods performed at baseline and after 6 cycles of neoadjuvant chemotherapy (NACT) are in agreement with histological findings from pre-treatment biopsy and post-treatment surgically excised tissue. MR methods will be performed at baseline (pre-treatment) and after the 1st, 3rd and 6th (post-treatment) cycles of NACT treatment. The investigators hypothesise that specific physiological changes detected through MR methods are a manifestation of tumour response to NACT confirmed by histology and radiological assessment (Hypothesis 1). The investigators further hypothesise that early sensitivity to physiological changes manifesting from tumour response to NACT can be revealed by MR measurements after the first and third cycle of treatment (Hypothesis 2).

Research Question 1: Is there a difference in physiological parameters revealed by MR measurements at baseline and after completion of NACT?

Research Question 2: Do the physiological measurements at the completion of NACT from MR measures agree with histological findings?

Research Question 3: Is there a difference between MR measurements at baseline and after the first and third cycle of NACT?

Research Question 4: Is there a difference in MR measurements at baseline, first and third cycle of NACT, between positive treatment responders and non-responders.

MR measurements will be compared against clinical and study specific results from histological analysis and radiological assessment of MRI, mammography and ultrasound measures of tumour treatment response. Information collected from a health questionnaire will supplement interpretation of the data.

To test the effects of NACT on specific aspects of tumour physiology, paired t-tests will be performed on MR measures of lactate concentration, lipid composition and diffusion parameters, between baseline and post-treatment assessments (Research Question 1).

To examine the relationship between MR measurements and histology, correlation analysis will be conducted between baseline and post-treatment assessments. MR measures will be correlated against corresponding percentage changes in histological findings between biopsy and tumour excision (Research Question 2).

To evaluate MR measures as early markers of NACT efficacy, paired t-tests will be carried out between MR measures at pre-treatment and post 1st and 3rd cycles of NACT treatment (Research Question 3), with independent group difference determined between responders and non-responders (Research Question 4).

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed invasive breast cancer undergoing neoadjuvant chemotherapy and surgery.

Exclusion Criteria:

* Condition to contradictive to MRI investigation with contrast agent (poor renal function, contrast agent allergy, metal implants or pace maker).
* Started hormone or chemotherapy treatment before recruitment.
* Undergoing treatment for concurrent cancer diagnosis.
* Marker coil contradictive to MRI investigation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Baseline: Water diffusion probability density function (Full-Width-At-Half-Maximum, FWHM, units of micrometre) | Scan at pre-treatment baseline (Prior to start of Cycle 1, each cycle is 21 days)
  The water diffusion probability density function will be quantified by the Full-Width-At-Half-Maximum with units of micrometre
Post Cycle 1: Water diffusion probability density function (Full-Width-At-Half-Maximum, FWHM, units of micrometre) | Scan at the end of Cycle 1 (Each cycle is 21 days)
  The water diffusion probability density function will be quantified by the Full-Width-At-Half-Maximum with units of micrometre
Post Cycle 3: Water diffusion probability density function (Full-Width-At-Half-Maximum, FWHM, units of micrometre) | Scan at the end of Cycle 3 (Each cycle is 21 days)
  The water diffusion probability density function will be quantified by the Full-Width-At-Half-Maximum with units of micrometre
Post Treatment: Water diffusion probability density function (Full-Width-At-Half-Maximum, FWHM, units of micrometre) | Scan at the end of Cycle 6 (Each cycle is 21 days)
  The water diffusion probability density function will be quantified by the Full-Width-At-Half-Maximum with units of micrometre
Baseline: Water diffusivity (units of mm^2 /s) | Scan at pre-treatment baseline (Prior to start of Cycle 1, each cycle is 21 days)
  Water diffusivity with units of mm^2 /s
Post Cycle 1: Water diffusivity (units of mm^2 /s) | Scan at the end of Cycle 1 (Each cycle is 21 days)
  Water diffusivity with units of mm^2 /s
Post Cycle 3: Water diffusivity (units of mm^2 /s) | Scan at the end of Cycle 3 (Each cycle is 21 days)
  Water diffusivity with units of mm^2 /s
Post Treatment: Water diffusivity (units of mm^2 /s) | Scan at the end of Cycle 6 (Each cycle is 21 days)
  Water diffusivity with units of mm^2 /s
Baseline: Lactate Concentration (units of mM) | Scan at pre-treatment baseline (Prior to start of Cycle 1, each cycle is 21 days)
  Lactate concentration with units of mM
Post Cycle 1: Lactate Concentration (units of mM) | Scan at the end of Cycle 1 (Each cycle is 21 days)
  Lactate concentration with units of mM
Post Cycle 3: Lactate Concentration (units of mM) | Scan at the end of Cycle 3 (Each cycle is 21 days)
  Lactate concentration with units of mM
Post Treatment: Lactate Concentration (units of mM) | Scan at the end of Cycle 6 (Each cycle is 21 days)
  Lactate concentration with units of mM
Baseline: Lipid Peak Volume Ratio (Ratio Units) | Scan at pre-treatment baseline (Prior to start of Cycle 1, each cycle is 21 days)
  Lipid peak volume ratio value with units of ratio
Post Cycle 1: Lipid Peak Volume Ratio (Ratio Units) | Scan at the end of Cycle 1 (Each cycle is 21 days)
  Lipid peak volume ratio value with units of ratio
Post Cycle 3: Lipid Peak Volume Ratio (Ratio Units) | Scan at the end of Cycle 3 (Each cycle is 21 days)
  Lipid peak volume ratio value with units of ratio
Post Treatment: Lipid Peak Volume Ratio (Ratio Units) | Scan at the end of Cycle 6 (Each cycle is 21 days)
  Lipid peak volume ratio value with units of ratio
Baseline: Fat Fraction (units of %) | Scan at pre-treatment baseline (Prior to start of Cycle 1, each cycle is 21 days)
  Fat Fraction with units of %
Post Cycle 1: Fat Fraction (units of %) | Scan at the end of Cycle 1 (Each cycle is 21 days)
  Fat Fraction with units of %
Post Cycle 3: Fat Fraction (units of %) | Scan at the end of Cycle 3 (Each cycle is 21 days)
  Fat Fraction with units of %
Post Treatment: Fat Fraction (units of %) | Scan at the end of Cycle 6 (Each cycle is 21 days)
  Fat Fraction with units of %

SECONDARY OUTCOMES:
Core Biopsy Tumour Tissue: Ki-67 Staining Percentage (units of %) | Pre-treatment baseline biopsy (Taken prior to start of Cycle 1, each cycle is 21 days). Assessed following completion of treatment cycles and the routine reporting of core biopsy and excised tissue samples.
  Ki-67 staining percentage with units of %, assessed on core biopsy tissue taken prior to start of treatment cycles.
Excised Tumour Tissue: Ki-67 Staining Percentage (units of %) | Post-treatment surgery excision (Post Cycle 6, each cycle is 21 days). Assessed following the completion of routine pathological reporting of the excised tissue.
  Ki-67 staining percentage with units of %, assessed on excised tissue taken from surgery following completion of treatment cycles.
Core Biopsy Tumour Tissue: Serotonin Staining Score (arbitrary units) | Pre-treatment baseline biopsy (Taken prior to start of Cycle 1, each cycle is 21 days). Assessed following completion of treatment cycles and the routine reporting of core biopsy and excised tissue samples.
  Serotonin staining score with arbitrary units (multiplication of staining percentage and stain intensity scored 1 - 3), assessed on core biopsy tissue taken prior to start of treatment cycles.
Excised Tumour Tissue: Serotonin Staining Score (arbitrary units) | Post-treatment surgery excision (Post Cycle 6, each cycle is 21 days). Assessed following the completion of routine pathological reporting of the excised tissue.
  Serotonin staining score with arbitrary units (multiplication of staining percentage and stain intensity scored 1 - 3), assessed on excised tissue taken from surgery following completion of treatment cycles.
Core Biopsy Tumour Tissue: Cellularity (units of %) | Pre-treatment baseline biopsy (Taken prior to start of Cycle 1, each cycle is 21 days). Assessed following completion of treatment cycles and the routine reporting of core biopsy and excised tissue samples.
  Cellularity with units of %, assessed on core biopsy taken prior to start of treatment cycles.
Excised Tumour Tissue: Cellularity (units of %) | Post-treatment surgery excision (Post Cycle 6, each cycle is 21 days). Assessed following the completion of routine pathological reporting of the excised tissue.
  Cellularity with units of %, assessed on excised tissue taken from surgery following completion of treatment cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Jiabao He, PhD, Study Chair — University of Aberdeen; Nicholas Senn, MPhys, Principal Investigator — University of Aberdeen
Locations (1):
- NHS Grampian, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MC, Newman LA. Management of patients with locally advanced breast cancer. Surg Clin North Am. 2007 Apr;87(2):379-98, ix. doi: 10.1016/j.suc.2007.01.012. PMID 17498533
- [Background] Luangdilok S, Samarnthai N, Korphaisarn K. Association between Pathological Complete Response and Outcome Following Neoadjuvant Chemotherapy in Locally Advanced Breast Cancer Patients. J Breast Cancer. 2014 Dec;17(4):376-85. doi: 10.4048/jbc.2014.17.4.376. Epub 2014 Dec 26. PMID 25548587
- [Background] Graham LJ, Shupe MP, Schneble EJ, Flynt FL, Clemenshaw MN, Kirkpatrick AD, Gallagher C, Nissan A, Henry L, Stojadinovic A, Peoples GE, Shumway NM. Current approaches and challenges in monitoring treatment responses in breast cancer. J Cancer. 2014 Jan 5;5(1):58-68. doi: 10.7150/jca.7047. PMID 24396498
- [Background] Danishad KK, Sharma U, Sah RG, Seenu V, Parshad R, Jagannathan NR. Assessment of therapeutic response of locally advanced breast cancer (LABC) patients undergoing neoadjuvant chemotherapy (NACT) monitored using sequential magnetic resonance spectroscopic imaging (MRSI). NMR Biomed. 2010 Apr;23(3):233-41. doi: 10.1002/nbm.1436. PMID 20175134
- [Background] Woodhams R, Kakita S, Hata H, Iwabuchi K, Kuranami M, Gautam S, Hatabu H, Kan S, Mountford C. Identification of residual breast carcinoma following neoadjuvant chemotherapy: diffusion-weighted imaging--comparison with contrast-enhanced MR imaging and pathologic findings. Radiology. 2010 Feb;254(2):357-66. doi: 10.1148/radiol.2542090405. PMID 20093508
- [Background] Walenta S, Mueller-Klieser WF. Lactate: mirror and motor of tumor malignancy. Semin Radiat Oncol. 2004 Jul;14(3):267-74. doi: 10.1016/j.semradonc.2004.04.004. PMID 15254870
- [Background] Carmona-Fontaine C, Bucci V, Akkari L, Deforet M, Joyce JA, Xavier JB. Emergence of spatial structure in the tumor microenvironment due to the Warburg effect. Proc Natl Acad Sci U S A. 2013 Nov 26;110(48):19402-7. doi: 10.1073/pnas.1311939110. Epub 2013 Nov 11. PMID 24218566
- [Background] Bolan PJ, Meisamy S, Baker EH, Lin J, Emory T, Nelson M, Everson LI, Yee D, Garwood M. In vivo quantification of choline compounds in the breast with 1H MR spectroscopy. Magn Reson Med. 2003 Dec;50(6):1134-43. doi: 10.1002/mrm.10654. PMID 14648561
- [Background] Baik HM, Su MY, Yu H, Mehta R, Nalcioglu O. Quantification of choline-containing compounds in malignant breast tumors by 1H MR spectroscopy using water as an internal reference at 1.5 T. MAGMA. 2006 May;19(2):96-104. doi: 10.1007/s10334-006-0032-4. Epub 2006 May 9. PMID 16779565
- [Background] He Q, Shkarin P, Hooley RJ, Lannin DR, Weinreb JC, Bossuyt VI. In vivo MR spectroscopic imaging of polyunsaturated fatty acids (PUFA) in healthy and cancerous breast tissues by selective multiple-quantum coherence transfer (Sel-MQC): a preliminary study. Magn Reson Med. 2007 Dec;58(6):1079-85. doi: 10.1002/mrm.21335. PMID 17969083
- [Background] Naressi A, Couturier C, Castang I, de Beer R, Graveron-Demilly D. Java-based graphical user interface for MRUI, a software package for quantitation of in vivo/medical magnetic resonance spectroscopy signals. Comput Biol Med. 2001 Jul;31(4):269-86. doi: 10.1016/s0010-4825(01)00006-3. PMID 11334636
- [Background] Yamada I, Hikishima K, Miyasaka N, Tokairin Y, Ito E, Kawano T, Kobayashi D, Eishi Y, Okano H. Esophageal carcinoma: Evaluation with q-space diffusion-weighted MR imaging ex vivo. Magn Reson Med. 2015 Jun;73(6):2262-73. doi: 10.1002/mrm.25334. Epub 2014 Jun 19. PMID 24947492
- [Derived] Cheung SM, Wu WS, Senn N, Sharma R, McGoldrick T, Gagliardi T, Husain E, Masannat Y, He J. Towards detection of early response in neoadjuvant chemotherapy of breast cancer using Bayesian intravoxel incoherent motion. Front Oncol. 2023 Dec 6;13:1277556. doi: 10.3389/fonc.2023.1277556. eCollection 2023. PMID 38125950